CLINICAL TRIAL: NCT06817122
Title: Mechanistic Study of the "Let's Talk Tech" Dyadic Behavioral Intervention to Support Decision Making About Technology Use
Brief Title: The "Let's Talk Tech" Tool to Support Decision Making About Technology Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Clara Berridge, Associate Professor: School of Social Work, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00020570; 1P30AG086562-01 (NIH)
Record Dates: First submitted 2025-01-03; First posted 2025-02-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Dementia, Mild; Mild Cognitive Impairment (MCI)
Keywords: Let's Talk Tech; shared decision aid; technology decision making; advance care planning; dyadic intervention
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Let's Talk Tech intervention (Experimental): The intervention group will complete the single use self-administered Let's Talk Tech intervention together as a dyad.
  Interventions: Behavioral: Let's Talk Tech
- Usual care (No Intervention): This control group will receive usual care, which means they will complete no intervention.

INTERVENTIONS:
Behavioral: Let's Talk Tech — Let's Talk Tech is a self-administered dyadic education and communication tool delivered as a web application to support shared decision making about technology use.
  Arms: Let's Talk Tech intervention

SUMMARY:
The goal of this research is to educate people about different technologies to support care at home when someone is experiencing memory difficulties. "Let's Talk Tech" is a new tool to educate people about technologies commonly used to support care and monitor safety, and help families talk about their feelings about them to understand each other's perspectives. The goal of this clinical trial is to learn if "Let's Talk Tech" helps people feel more prepared to make decisions about technologies.

Researchers will compare Let's Talk Tech to usual care (no intervention) to see if Let's Talk Tech increases peoples' preparedness and confidence to make decisions about technologies.

Participants will:

* Use the Let's Talk Tech web application together with their study partner that takes up to an hour or do nothing.
* Complete three surveys. The second survey will be taken within 2 weeks of the first and the last survey will be taken 3 months after the first.

DETAILED DESCRIPTION:
The goal of this research is to help families understand digital health technology options to support dementia care at home so they can negotiate immediate decisions and future use in an informed way. This is a mechanism-focused trial of Let's Talk Tech (LTT), a single-use, self-administered intervention in the form of a web application. It targets education and interpersonal communication processes to enable informed decision making and planning for technology use that relieves care partners of the burden of making decisions without awareness of the person's preferences. Participants are people living with mild Alzheimer's disease (AD) and AD-related dementias (PLWD) or mild cognitive impairment (MCI) and a care partner. The 120 enrolled dyads (60 per study group) will be randomly assigned to receive either the intervention or usual care control. The intervention is self-administered. All participants will complete measures at baseline, at post-test (2 weeks) and 3 months later. Aim 1 will test if LTT compared with usual care improves the hypothesized mechanisms of change that are care partners' technology awareness, understanding, communication satisfaction, and intention to honor the PLWD/MCI's preferences, as well as both care partner- and PLWD/MCI-reported dyadic alignment. Aim 2 will examine if and how those hypothesized mechanisms of change improve the post-test and 3-month primary outcomes of care partner preparedness and decisional conflict, and secondary outcomes of PLWD/MCI and care partner sharing of technology preferences beyond the dyad and their confidence that PLWD/MCI's preferences will be honored. Exploratory Aim 3 will examine how, with whom, and for what purpose dyad members share technology preferences and explore factors that vary for those who shared with providers vs. family/friends, with the hope of learning how to expand the reach of this intervention to activate dyads' entire care networks.

ELIGIBILITY:
Inclusion Criteria for Patients:

* have mild cognitive impairment (MCI) or mild dementia
* age 55 or older
* able to understand and speak English

Inclusion Criteria for Co-participants:

* be identified by the patient as their primary support person
* age 18 or older
* able to understand and speak English
* able to complete LTT together with their study partner at the same time

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Preparedness to make technology decisions | baseline, 2-week post-test and 3 months
  Participant rates on a 5-point Likert scale [1="Strongly agree" to 5="Strongly disagree"] how much they agree with the statement that they feel prepared to make decisions about technology use for their study partner.
Decisional Conflict Scale | baseline, 2-week post-test and 3 months
  The Decisional Conflict Scale is a 16-item scale with 5 response categories [0= "Strongly agree" to 4="Strongly disagree"]. Higher scores reflect higher decisional conflict in decision making.
Technology awareness | baseline and 2-week post-test
  Participant rates on a 5-point Likert scale [1="Very aware" to 5="Very unaware"] how aware they are about technologies available to support their partner's care and safety.
Technology understanding | baseline and 2-week post-test
  4 items assess perceived understanding of each of 4 technologies featured in the intervention [1="Not at all" to 5="Completely"].
Perception of PLWD/MCI's technology understanding | baseline and 2-week post-test
  4 items assess care partner's perception of how well their study partner understands of each of 4 technologies featured in the intervention [1="Not at all" to 5="Completely"].
Satisfaction with dyadic communication about technology | baseline and 2-week post-test
  Participant rates on a 5-point Likert scale [1="Very satisfied" to 5="Very dissatisfied"] how satisfied they are with their discussion with their study partner about using technology to support their care or safety.
Intention to honor preferences | baseline and 2-week post-test
  Participant rates on a 5-point Likert scale [1="Very likely" to 5="Very unlikely"] how likely they are to honor their partner's preferences for how technology is used in their care.
Dyadic alignment about technology use | baseline and 2-week post-test
  Participant is asked how much they agree with their partner about using technologies to support their care [1="Not at all" to 5="Completely"].

SECONDARY OUTCOMES:
Shared technology preferences | baseline, 2-week post-test and 3 months
  Participant answer yes or no if they have ever shared the PLWD/MCI's preferences about technologies to support their care with anyone else.
Confidence preferences will be honored | baseline, 2-week post-test and 3 months
  Participant rates on a 5-point Likert scale [1=Strongly agree to 5=Strongly disagree] about their belief the PLWD/MCI's choices about these technologies will be honored.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Berridge, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No